CLINICAL TRIAL: NCT04748406
Title: Comparison of Peloidotherapy and Extracorporeal Shock Wave Therapy Efficiency in Patients With Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Hasan Koru, assistant doctor, Konya Meram State Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KonyaTRH1
Record Dates: First submitted 2021-01-16; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Lateral Epicondylitis
Keywords: Extracorporeal Shock Wave Therapy; Peloidotherapy
MeSH Terms: conditions — Tennis Elbow | interventions — Extracorporeal Shockwave Therapy; Mud Therapy

STUDY DESIGN:
Intervention Model Description: The study was designed as prospective, case-control and hospital-based.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peloid Therapy (Active Comparator): Group 1 (n = 35) will be given 15 sessions of peloid therapy + cold application + home exercise program for 3 weeks, 5 days a week(16).
  Interventions: Other: Peloid therapy; Other: Home Workout Program; Other: Cold application
- ESWT(Extracorporeal Shock Wave Therapy) (Active Comparator): Group 2 (n = 35) will be applied 1 session per week for 3 weeks, 3 sessions of ESWT (1.8 bar, 10.0 Hz, 2000 beats) + cold application + home exercise program will be applied(4).
  Interventions: Device: Extracorporeal Shock Wave Therapy(ESWT); Other: Home Workout Program; Other: Cold application

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy(ESWT) — Group 2 (n = 35) will be applied 1 session per week for 3 weeks, 3 sessions of ESWT (1.8 bar, 10.0 Hz, 2000 beats) + cold application + home exercise program will be applied.
  Arms: ESWT(Extracorporeal Shock Wave Therapy)
Other: Peloid therapy — Group 1 (n = 35) will be given 15 sessions of peloid therapy + cold application + home exercise program for 3 weeks, 5 days a week
  Arms: Peloid Therapy
Other: Home Workout Program — Patients will be given a home exercise program consisting of eccentric strengthening exercises and stretching exercises, which are planned to increase resistance every week. The patients will be taught strengthening exercises for forearm pronation-supination with wrist extensors and a home exercise program will be started 3 sets of 10 repetitions per day.
Other: Cold application — At the beginning of each treatment, gel ice packs are wrapped with a moist towel and placed around the elbow joint for 15 minutes. will be applied.

SUMMARY:
Investigator could not find a study comparing ESWT(Extracorporeal Shock Wave Therapy) and Peloidotherapy methods in the treatment of lateral epicondylitis in the literature. Therefore, in this study, it was planned to investigate the difference in effectiveness between Peloidotherapy and ESWT in the treatment of Lateral Epicondylitis.

DETAILED DESCRIPTION:
The frequency of lateral epicondylitis (LE), one of the most common causes of elbow pain, has been reported to be 1-3%. It is usually seen between the ages of 40-50 and the dominant side is more frequently affected. The most common cause of elbow lateral pain in adults is LE (1,2). Pain that occurs in LE and radiates to the humerus and forearm is characteristic of this disease. (3). The diagnosis of lateral epicondylitis is usually made clinically. Dorsiflexion of the wrist against resistance, pressure on the lateral epicondyle and firm grip of an object causes pain radiating to the forearm. (4). With appropriate conservative treatments, 75-90% relief has been reported in patients with LE (1). Chronic symptoms develop in 5-10% of the patients. Various treatments have been tried to reduce the pain of the patient and increase the functions in LE, which restricts daily life activities. Although many treatment methods are used in the treatment of LE disease, it is controversial which is the most effective method. Extracorporeal Shock Wave therapy (ESWT), peloidotherapy, NSAID, corticosteroid injection, cold application, fascia loosening, electrotherapy applications, kinesio band, iontophoresis, splint, orthosis, acapuntur, ultrasound therapy, deep friction massage, exercise, manipulation, mobilization, laser, Botulinum toxin injection, tenotomy, and autologous blood injections are among the recommended treatments (4-9). Although there are so many different treatment methods in the treatment of lateral epicondylitis, there is no consensus on which one is the most effective and successful.

Peloids (medicinal mud) are organic or inorganic substances formed as a result of geological and / or biological events. They can be found in nature as fine particles, or they are made into small, fine particles by some pre-preparation processes. (10). Peloidotherapy is a special balneotherapy method made with natural muds (11). It is especially used in the treatment of diseases such as degenerative joint diseases, soft tissue rheumatism, lumbar discopathy, cervical discopathy, chronic back and neck pain, joint pain. Scientific studies on peloid treatment both in Turkey and abroad have shown that patients have reduced pain (12), improved physical functions, increased quality of life, and decreased pain medication use (12-15). A recent study demonstrated the effectiveness of peloidotherapy in LE. (16). Ökmen et al. In this study, the effectiveness of peloidotherapy and elbow bandage in the treatment of LE was compared. (16). This study remains the only one investigating the effectiveness of peloidotherapy in the treatment of LE.

Shock wave therapy (extracorporeal shock wave therapy, Extracorporeal Shock Wave Therapy-ESWT) is a new orthopedic treatment method based on focusing high amplitude sound waves on the desired area of the body and providing treatment there. (17). ESWT creates a cavitation effect in deep tissue by creating capillary microrupture, chemical mediator leakage, and neovascularization in damaged tissue with low or high energy options (18). Successful results have been reported with ESWT treatment in 48-73% of cases with recurrent LE with non-surgical methods (19). Due to its non-invasive nature and low complication rates, the use of ESWT in LE treatment is gradually increasing (20). Some authors state that ESWT has lateral LE effect (20). Some authors reported that ESWT is not in the treatment of LE (21).

Investigator did not find a study comparing ESWT and Peloidotherapy methods in the treatment of LE in the literature. In this thesis, our aim is to compare the effectiveness of peloidotherapy and ESWT methods used in the treatment of LE with a prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with elbow pain and are diagnosed with unilateral LE due to the presence of pain by pressing on the epicondyle in physical examination, wrist extension against resistance and during stretching of the wrist extensors, who have elbow pain for at least 3 months and between the ages of 18-65 will be accepted to the study.

Exclusion Criteria

* Those with communication problems
* A history of cervical and shoulder problems
* History of injection, surgery, physical therapy in the elbow area in the last 6 months
* Having had ESWT treatment in the elbow area before
* History of elbow problems other than LE
* Elbow osteoarthritis, previous elbow fracture history
* A history of polyneuropathy,
* Those with a history of uncontrolled systemic disease (cardiovascular, pulmonary, hepatic, renal, hematologic ..),
* Those with a history of systemic endocrine disease (DM, hyperthyroidism ..),
* Major psychiatric illness
* History of rheumatic diseases such as fibromyalgia, polymyalgiaromatica, ankylosing spondylitis, rheumatoid arthritis
* Those who use bleeding disorders and anticoagulants
* Neurological deficit
* Malignancy
* Those with a history of pacemakers were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Descriptive Characteristics of Patients | All evaluations will be applied one time by the same investigator in both groups, at the beginning of the treatment.
  Patients were questioned about age, gender, body mass index (BMI), education level, occupation, the extremity affected by the dominant, duration of complaints, previous treatments and when the last treatment was administered.
Evaluation of Grip Force Change | All evaluations will be applied three times by the same investigator in both groups, at the beginning of the treatment, in the 3rd week after the treatment, and on the 4th week after the end of the treatment.
  The grip strength of the hand is accepted as the most objective criterion of the functional integrity of the upper extremity. Hand grip strength also provides convenience and objectivity in evaluating the treatment. (26). It is known that hand grip strength measurements with the Jamar hand dynamometer, which is one of the methods used for this purpose, give reliable results (22, 26, 27). Jamar dynamometer will be used in hand grip strength measurements.
Evaluation of Subjective Pain Intensity Change | All evaluations will be applied three times by the same investigator in both groups, at the beginning of the treatment, in the 3rd week after the treatment, and on the 4th week after the end of the treatment.
  Pain interrogation using a 0-10 point Visual Analogue Scale (VAS) will be used to detect pain and disability caused by the disease. The questions were pain at rest, pain during straining, pain relief effectiveness, subjective work failure, difficulty in lifting 2 kg objects, inability during hobby activities and sleep disturbance. Patients were asked to answer each question as 0 (no pain or disability) 10 (worst possible pain or disability) on a scale of 0-10 cm. The total pain score, which is the sum of 7 different sub-scores, will be calculated for each patient. In addition to 0-10 point Visual Analogue Scale (VAS) was used to evaluate the severity of pain during maximum hand grip.
Treatment Satisfaction Level Change | All evaluations will be applied two times by the same investigator in both groups, in the 3rd week after the treatment, and on the 4th week after the end of the treatment.
  "Roles and Maudsley Scoring" will be used to measure the treatment satisfaction level of the patients. The "Roles and Maudsley Scoring" is a measure of whether patients with lateral epicondylitis benefit from treatment. It is scored between 1 and 4 points. 1 point indicates that satisfaction with treatment and benefit from treatment is high. As the score level increases, the level of satisfaction and benefit from treatment decreases. 4 points show that he did not benefit from the treatment at all and he was not satisfied.
Evaluation of Functionality Level Change | All evaluations will be applied three times by the same investigator in both groups, at the beginning of the treatment, in the 3rd week after the treatment, and on the 4th week after the end of the treatment.
  Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire; The field-specific outcome measurement DASH questionnaire has been developed to evaluate functional status and symptoms in musculoskeletal disorders occurring in the upper extremity.The DASH questionnaire consists of 3 parts. The first part consists of 30 questions; 21 questions assess the patient's difficulties during daily life activities, 5 questions evaluate symptoms (pain, activity-related pain, tingling, stiffness, weakness), and each of the remaining 4 questions assess social function, work, sleep and patient self-confidence.
Evaluation of Functionality Level Change | All evaluations will be applied three times by the same investigator in both groups, at the beginning of the treatment, in the 3rd week after the treatment, and on the 4th week after the end of the treatment.
  Patient-Rated Forearm Evaluation Questionnaire(PRFEQ), a Turkish validated scoring system, is designed to assess arm pain and functions over a 1-week period. It questions how much pain and difficulty you have had with your arm over the past week. Pain is assessed with 5 questions and functions with 10 questions. The subtitles of PRFEQ related to pain are scored between 0 (no pain) and 10 (worst possible pain) on a 0-10 cm VAS scale.
Evaluation of Quality of Life Change | All evaluations will be applied three times by the same investigator in both groups, at the beginning of the treatment, in the 3rd week after the treatment, and on the 4th week after the end of the treatment.
  The SF-36 (the MOS 36-item short-form health survey) Health Survey is a 36-question questionnaire consisting of 8 subgroups to measure the general quality of life. It is filled by the patient himself. It has eight subgroups (general health, physical function, physical condition, pain, life functions, social functions, emotional state, mental health) and 2 summary scales (mental health and physical health). It is scored between 0 and 100, with 0 reporting the worst health condition, 100 the best health condition.

CONTACTS AND LOCATIONS:
Overall Officials: hasan koru, Principal Investigator — assistant doctor
Locations (1):
- Konya Beyhekim Training and Research Hospital Physical Medicine and Rehabilitation Clinic, Selçuklu, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
1 year after publication in the journal under sci
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: April 2023 - April 2025
Access Criteria: 1 year after publication in the journal under sci

REFERENCES:
- [Background] 1.Barrington J, Hage W. Lateral epicondylitis (tenis elbow): nonoperative, open, or arthroscopic treatment?. Curr Opin Orthop 2003; 14: 291-295.
- [Background] 2.Chard MD. The Elbow. In Hochberg MC, Silman AJ, Smolen JS, Weinblatt ME, Weisman MH, editors. Rheumatology. 3rd ed. Mosby, London; 2003. p. 631-9.
- [Background] Shiri R, Viikari-Juntura E, Varonen H, Heliovaara M. Prevalence and determinants of lateral and medial epicondylitis: a population study. Am J Epidemiol. 2006 Dec 1;164(11):1065-74. doi: 10.1093/aje/kwj325. Epub 2006 Sep 12. PMID 16968862
- [Background] 4.Soner Akkurt, Ahmet Yılmaz, Tolga Saka. Lateral epikondilit tedavisinde ekstrakorporeal şok dalga tedavisi, fizyoterapi ve lokal steroid enjeksiyonunun karşılaştırılması Turk J Phys Med Rehab 2016;1(62):37-44.
- [Background] Derebery VJ, Devenport JN, Giang GM, Fogarty WT. The effects of splinting on outcomes for epicondylitis. Arch Phys Med Rehabil. 2005 Jun;86(6):1081-8. doi: 10.1016/j.apmr.2004.11.029. PMID 15954044
- [Background] 6. Ölmez N, Memiş A. Lateral Epikondilit Tedavisinde Kanıta Dayalı Veriler. Rewiev . Turkiye Klinikleri J Med Sci 2010;30(1)
- [Background] Foley AE. Tennis elbow. Am Fam Physician. 1993 Aug;48(2):281-8. PMID 8342481
- [Background] Wilson JJ, Best TM. Common overuse tendon problems: A review and recommendations for treatment. Am Fam Physician. 2005 Sep 1;72(5):811-8. PMID 16156339
- [Background] 9. Aydin A, Celepkolu T, Atiç R, Alemdar C, Aydin ZS, Cevik R. Effects of Extracorporeal Shock Wave Therapy On The Quality of Life And Pain in Patients With Lateral Epicondylitis. Euras J Fam Med 2018;7(1):29-36
- [Background] 10. Karagülle MZ. Balneoloji ve Kaplıca Tıbbı. İstanbul: Nobel Tıp Kitabevleri; 2002. s. 15-36.
- [Background] 11. Özer UN. Kaplıca Tedavisi. In: Tuna N, Eds. Romatizmal Hastalıklar. Ankara: Hacettepe Taş Kitapçılık; 1994. s. 229-42.
- [Background] Fioravanti A, Bacaro G, Giannitti C, Tenti S, Cheleschi S, Gui Delli GM, Pascarelli NA, Galeazzi M. One-year follow-up of mud-bath therapy in patients with bilateral knee osteoarthritis: a randomized, single-blind controlled trial. Int J Biometeorol. 2015 Sep;59(9):1333-43. doi: 10.1007/s00484-014-0943-0. Epub 2014 Dec 17. PMID 25516113
- [Background] Liu H, Zeng C, Gao SG, Yang T, Luo W, Li YS, Xiong YL, Sun JP, Lei GH. The effect of mud therapy on pain relief in patients with knee osteoarthritis: a meta-analysis of randomized controlled trials. J Int Med Res. 2013 Oct;41(5):1418-25. doi: 10.1177/0300060513488509. Epub 2013 Sep 5. PMID 24008567
- [Background] Espejo-Antunez L, Cardero-Duran MA, Garrido-Ardila EM, Torres-Piles S, Caro-Puertolas B. Clinical effectiveness of mud pack therapy in knee osteoarthritis. Rheumatology (Oxford). 2013 Apr;52(4):659-68. doi: 10.1093/rheumatology/kes322. Epub 2012 Dec 11. PMID 23236190
- [Background] Tefner IK, Gaal R, Koroknai A, Rathonyi A, Gati T, Monduk P, Kiss E, Kovacs C, Balint G, Bender T. The effect of Neydharting mud-pack therapy on knee osteoarthritis: a randomized, controlled, double-blind follow-up pilot study. Rheumatol Int. 2013 Oct;33(10):2569-76. doi: 10.1007/s00296-013-2776-2. Epub 2013 May 21. PMID 23689969
- [Background] Okmen BM, Eroksuz R, Altan L, Aksoy MK. Efficacy of peloid therapy in patients with chronic lateral epicondylitis: a randomized, controlled, single blind study. Int J Biometeorol. 2017 Nov;61(11):1965-1972. doi: 10.1007/s00484-017-1386-1. Epub 2017 Jun 15. PMID 28620677
- [Background] 17.İsmail Baloğlu, M. Hakan Özsoy, Hilmi Aydınok, Veli Lök. Ortopedi ve Travmatolojide Şok Dalga Tedavisi. TOTBİD (Türk Ortopedi ve Travmatoloji Birliği Derneği) Dergisi. 2005 • Cilt: 4 Sayı: 1-2.
- [Background] 18. Hossain M, Makwana N. "Not Plantar Fasciitis": the differential diagnosis and management of heel pain syndrome. Orthop Trauma. 2011;25:198-206
- [Background] Ogden JA, Alvarez RG, Levitt R, Marlow M. Shock wave therapy (Orthotripsy) in musculoskeletal disorders. Clin Orthop Relat Res. 2001 Jun;(387):22-40. doi: 10.1097/00003086-200106000-00005. PMID 11400888
- [Background] Bayram K, Yesil H, Dogan E. Efficacy of extracorporeal shock wave therapy in the treatment of lateral epicondylitis. North Clin Istanb. 2014 Aug 3;1(1):33-38. doi: 10.14744/nci.2014.77487. eCollection 2014. PMID 28058299
- [Background] Melikyan EY, Shahin E, Miles J, Bainbridge LC. Extracorporeal shock-wave treatment for tennis elbow. A randomised double-blind study. J Bone Joint Surg Br. 2003 Aug;85(6):852-5. PMID 12931804
- [Background] Schmidt RT, Toews JV. Grip strength as measured by the Jamar dynamometer. Arch Phys Med Rehabil. 1970 Jun;51(6):321-7. No abstract available. PMID 5423802
- [Background] 23. Düger T, Yakut E, Öksüz Ç, Yörükan S, Bilgütay BS, Ayhan Ç, Leblebicioğlu G, Kayıhan H, Kırdı N, Yakut Y, Güler Ç. Kol, Omuz ve El Sorunları (Disabilities of the Arm, Shoulder and Hand - DASH) Anketi Türkçe uyarlamasının güvenirliği ve geçerliği. Fizyoterapi Rehabilitasyon. 2006; 17(3):99-107.
- [Background] Altan L, Ercan I, Konur S. Reliability and validity of Turkish version of the patient rated tennis elbow evaluation. Rheumatol Int. 2010 Jun;30(8):1049-54. doi: 10.1007/s00296-009-1101-6. Epub 2009 Aug 26. PMID 19707766
- [Background] 25. Koçyiğit H. Aydemir Ö, Fişek G. Kısa form-36(KF-36)'nın Türkçe versiyonunun güvenirliliği ve geçerliliği. İlaç ve Tedavi Dergisi.1999;12:102-106.
- [Background] Balogun JA, Akomolafe CT, Amusa LO. Grip strength: effects of testing posture and elbow position. Arch Phys Med Rehabil. 1991 Apr;72(5):280-3. PMID 2009042
- [Background] 27. Üncel NA, Ceceli E, Durukan BP, Öken Ö, Erdem HR. El kavrama gücüne cinsiyet ve el dominansının etkisinin değerlendirilmesi. Romatizma, Cilt: 17, Sayı: 1, 2002.
- [Background] Trampisch US, Franke J, Jedamzik N, Hinrichs T, Platen P. Optimal Jamar dynamometer handle position to assess maximal isometric hand grip strength in epidemiological studies. J Hand Surg Am. 2012 Nov;37(11):2368-73. doi: 10.1016/j.jhsa.2012.08.014. PMID 23101534
- [Background] Amaral JF, Mancini M, Novo Junior JM. Comparison of three hand dynamometers in relation to the accuracy and precision of the measurements. Rev Bras Fisioter. 2012 Jun;16(3):216-24. doi: 10.1590/s1413-35552012000300007. PMID 22801514
- [Background] 30. Feneis H. Sistematik Resimli Anatomi Sözlüğü (Çev. Ed: Yıldırım M) s. 90-92, Nobel Yüce, İstanbul, 1997.
- [Background] Pienimaki TT, Siira PT, Vanharanta H. Chronic medial and lateral epicondylitis: a comparison of pain, disability, and function. Arch Phys Med Rehabil. 2002 Mar;83(3):317-21. doi: 10.1053/apmr.2002.29620. PMID 11887110
- [Background] Roles NC, Maudsley RH. Radial tunnel syndrome: resistant tennis elbow as a nerve entrapment. J Bone Joint Surg Br. 1972 Aug;54(3):499-508. No abstract available. PMID 4340924
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Derived] Koru H, Yilmaz H, Yilmaz R, Karpuz S. Comparison of the efficiency of peloidotherapy and extracorporeal shock wave therapies in patients diagnosed with lateral epicondylitis: a prospective, randomized, controlled study. Int J Biometeorol. 2024 Jan;68(1):101-108. doi: 10.1007/s00484-023-02574-5. Epub 2023 Nov 7. PMID 37934301